CLINICAL TRIAL: NCT06734208
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Cohort Study to Evaluate the Pharmacokinetics of Divarasib in Subjects With Impaired Hepatic Function
Brief Title: A Study to Evaluate the Pharmacokinetics of Divarasib in Healthy Participants and Participants With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP45713
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants will receive a single oral dose of Divarasib on Day 1.
  Interventions: Drug: Divarasib
- Cohort 2 (Experimental): Participants will receive a single oral dose of Divarasib on Day 1.
  Interventions: Drug: Divarasib
- Cohort 3 (Experimental): Participants will receive a single oral dose of Divarasib on Day 1.
  Interventions: Drug: Divarasib
- Cohort 4 (Experimental): Participants will receive a single oral dose of Divarasib on Day 1.
  Interventions: Drug: Divarasib

INTERVENTIONS:
Drug: Divarasib — Divarasib will be administered as a single oral dose as specified for the respective cohort.

SUMMARY:
This is a phase 1, open-label, single-dose, parallel-cohort study to determine the pharmacokinetics (PK) of divarasib in healthy participants and participants with varying degrees of hepatic impairment, as defined by Child-Pugh classification.

ELIGIBILITY:
Key Inclusion Criteria

* Males or females of non-childbearing potential
* Within body mass index (BMI) range of 18.0 to 45.0 kg/m2

Participants with Hepatic Impairment

* Considered to have mild, moderate, or severe hepatic impairment by Child-Pugh Score classification and has been clinically stable for at least 1 month prior to Screening
* Chronic (>6 months), stable hepatic insufficiency with features of cirrhosis due to any etiology. Participants must also remain stable throughout the Screening period

Key Exclusion Criteria

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator

Participants with Hepatic Impairment

* Have a QTcF >480 msec for males and >490 msec for females at Screening or Check-in. If any parameter is out of range, the ECG may be repeated for confirmation
* Any evidence of progressive liver disease that has worsened or is worsening, as determined by the investigator, within 1 month prior to Screening
* Demonstrated evidence of hepatorenal syndrome
* Ascites requiring paracentesis or other intervention up to 3 days prior to the study
* Hepatic encephalopathy Grade 2 or above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Divarasib | Day 1 to Day 7
Maximum Observed Concentration (Cmax) of Divarasib | Day 1 to Day 7
Area Under the Concentration-time Curve from Hour 0 to the last measurable concentration (AUC0-t) of Divarasib | Day 1 to Day 7
Area Under the Concentration-time Curve Extrapolated to Infinity (AUC0-inf) of Divarasib | Day 1 to Day 7

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Panax Clinical Research, LLC, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No